CLINICAL TRIAL: NCT01841749
Title: Management of Ductal Carcinoma in Situ (DCIS) or Pure Micro-invasive (DCIS-MI) Extended Breast, Axillary Node Sentinel Site (GAS) When the Diagnosis is Made by Biopsy and Treatment by Mastectomy Immediately. Descriptive Study
Brief Title: Management of Ductal Carcinoma in Situ or Pure Micro-invasive Extended Breast
Acronym: CINNAMOME
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Other Study IDs: IB2007-40
Record Dates: First submitted 2012-11-05; First posted 2013-04-26 (Estimated); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Intraductal Carcinoma and Lobular Carcinoma in Situ
Keywords: Breast cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy; Mastectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Surgery: sentinel node biopsy and mastectomy
  Interventions: Procedure: sentinel node biopsy and mastectomy

INTERVENTIONS:
Procedure: sentinel node biopsy and mastectomy — sentinel node biopsy and mastectomy

SUMMARY:
When invasive components are discovered at mastectomy for vacuum-assisted biopsy (VAB)-diagnosed ductal carcinoma in situ (DCIS), the only option available is axillary lymph node dissection (ALND). The aim of this prospective multicenter trial was to determine the benefit of performing upfront sentinel lymph node (SLN) biopsy for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years.
* Preoperative histological diagnosis obtained by biopsy
* Ductal carcinoma in situ (DCIS) or pure micro-invasive (DCIS-MI)
* Indication of mastectomy
* Patient signed informed consent

Exclusion Criteria:

* Age < 18 years
* Infiltrating ductal carcinoma (TCC) diagnosed on biopsy
* Pure DCIS diagnosed by lumpectomy
* DCIS can take a conservative treatment
* Mastectomy chosen by the patient
* History of breast carcinoma in situ or invasive ipsilateral
* Prior radiotherapy to the ipsilateral breast
* History of axillary lateral homo
* Patient who for reasons psychological, social, family or geographical could not be treated or monitored regularly according to the criteria of the study
* Patient deprived of liberty or under guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were recruited from 14 participating French comprehensive cancer centers.
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: TUNON DE LARA Christine, MD, Study Chair — Institut Bergonié
Locations (1):
- Institut Bergonié, Bordeaux, Aquitaine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tunon-de-Lara C, Chauvet MP, Baranzelli MC, Baron M, Piquenot J, Le-Bouedec G, Penault-Llorca F, Garbay JR, Blanchot J, Mollard J, Maisongrosse V, Mathoulin-Pelissier S, MacGrogan G. The Role of Sentinel Lymph Node Biopsy and Factors Associated with Invasion in Extensive DCIS of the Breast Treated by Mastectomy: The Cinnamome Prospective Multicenter Study. Ann Surg Oncol. 2015 Nov;22(12):3853-60. doi: 10.1245/s10434-015-4476-5. Epub 2015 Mar 17. PMID 25777085

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Surgery
Started | 228
Completed | 227
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Surgery
Number analyzed (Participants) | 228
Age, Continuous [Median (Full Range); unit: years] | 52 [24 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 228
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 228

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Women Who Benefited of Performing Upfront Sentinel Lymph Node (SLN) Biopsy Ductal Carcinoma in Situ
Description: Women who benefited of performing upfront sentinel lymph node (SLN) biopsy are women for whom unecessary axillary lymph node dissection (ALND) was avoided.
  The proportion of women who benefited of performing upfront sentinel lymph node (SLN) biopsy is calculated as :
  * numerator : number of patients with negative SLNs
  * denominator : total number of patients with mastectomy-diagnosed DCIS with microinvasion (mDCIS-MI) or mastectomy-diagnosed DCIS with associated invasive carcinoma (mDCIS-IDC).
Time Frame: at surgery
Population: Women with mastectomy-diagnosed DCIS with microinvasion (mDCIS-MI) or mastectomy-diagnosed DCIS with associated invasive carcinoma (mDCIS-IDC).
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery
Number analyzed (Participants) | 76
Participants | 51

2. Secondary Outcome: Discordance Rate Between Vacuum-assisted Biopsy (VAB) and Mastectomy
Description: Numerator : number of patients with discordant results between VAB and mastectomy Denominator : total number of patients
Time Frame: at surgery
Population: Women with vacuum-assisted biopsy (VAB) diasgnosis available and mastectomy diagnosis available
Measure: Count of Participants; unit: Participants
Arm/Group | Surgery
Number analyzed (Participants) | 196
Participants | 76

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed for this prospective observational study
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed for this prospective observational study
Arm/Group | Surgery
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes